CLINICAL TRIAL: NCT06389448
Title: Comparison of Probe-based Confocal Laser Endomicroscopy and Traditional Endoscopic Biopsies in the Diagnosis of Gastric Cancer and Precancerous Lesions: a Prospective Multicenter Comparative Study
Brief Title: Comparison of pCLE and EB in Gastric Lesion Diagnosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Cheng, professor, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: pCLE vs EB 2024tj
Record Dates: First submitted 2024-04-22; First posted 2024-04-29 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Low Grade Intraepithelial Neoplasia; High Grade Intraepithelial Neoplasia; Early Gastric Cancer; Gastric Intraepithelial Neoplasia
Keywords: confocal laser endomicroscopy; endoscopic biopsy; Intraepithelial Neoplasia; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma in Situ

STUDY DESIGN:
Intervention Model Description: Participants undergo pCLE after pre-ESD assessment and before ESD resection.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pCLE-gastr (Other): pCLE will be used to acquire the images from the gastric tissue of the participants after preoperative fluorescein sodium allergy test (negative) and pre-ESD assessment，and before ESD resection.
  Interventions: Device: pCLE-gastr

INTERVENTIONS:
Device: pCLE-gastr — After identifying the location of the lesion through white light endoscopy, the pCLE operation is performed to acquire images from the specific gastric lesions, and finally the ESD routine is performed.

SUMMARY:
This is a prospective multicenter comparative study, aiming to compare probe-based confocal laser endomicroscopy (pCLE) and endoscopic biopsies in the diagnosis of the whole specific gastric lesion especially for distinguishing low grade intraepithelial neoplasia (LGIN) from high grade intraepithelial neoplasia (HGIN) and create an endoscopic image database for the follow-up research.

DETAILED DESCRIPTION:
Traditional endoscopic biopsies can only obtain limited tissues from the whole lesion and is invasive, while probe-based confocal laser endomicroscopy (pCLE) can obtain images at a cellular level of the entire lesion area in real time and non-invasively. There were only single-center and small-sample previous researches for comparing the diagnostic accuracy of CLE and traditional biopsy in the entire gastric lesions, and they did not distinguish gastric low grade intraepithelial neoplasia (LGIN) from high grade intraepithelial neoplasia (HGIN). Thus, this study aims to further verify whether pCLE or pCLE combined with biopsy can improve the diagnostic accuracy of the overall lesion and reduce the histological upstaging rate of gastric LGIN after endoscopic submucosal dissection (ESD) by using large sample data and a new pCLE classification method, so as to achieve better guidance of clinical treatment. While verifying the diagnostic efficacy of pCLE, the data of the participants will be collected and collated, and an endoscopic image database will be constructed for the follow-up research.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old and under 75 years old;
* Patients with pathological diagnosis of LGIN, HGIN or early gastric cancer after conventional endoscopy biopsy, whose lesion has clear boundaries under endoscopic observation and is to be admitted for ESD surgery;
* Patients who meet the indications for endoscopic resection of early gastric cancer, or LGIN patients who intend to undergo ESD surgery;
* Patients who are able to provide pathological specimens/sections of previous endoscopic biopsy (in principle, it should be a case of this center).

Exclusion Criteria:

* Patients with advanced gastric cancer or previous gastrectomy;
* Patients with severe cardiopulmonary dysfunction, liver cirrhosis, renal dysfunction, acute gastrointestinal bleeding, esophageal-gastro varices, and coagulation disorders;
* Patients who have a positive result in the fluorescein sodium allergy test;
* Pregnant and lactating women;
* Patients who have psychiatric disorders and are unable to cooperate with endoscopy or sign informed consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of pCLE and endoscopic biopsy in diagnosing the whole gastric lesion | immediatly after the diagnostic result of biopsy, ESD and pCLE is available，or admission up to 2 months
  Using the pathological diagnostic result as the criteria, the accuracy, sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) will be used to evaluate the diagnostic efficacy in diagnosing LGIN, HGIN and early gastric cancer.

SECONDARY OUTCOMES:
The histological upstaging rate of pCLE and endoscopic biopsy in diagnosing the whole gastric lesion | immediatly after the diagnostic result of biopsy, ESD and pCLE is available，or admission up to 2 months
  Using the pathological diagnostic result as the ending, the histological upstaging rate from endoscopic biopsy or pCLE will be used to evaluate the diagnostic efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China